CLINICAL TRIAL: NCT05437003
Title: A Cross-Sectional Study to Evaluate the Correlation Between Oculometric Measures and MDS-UPDRS in Patients With Idiopathic Parkinson's Disease (PD) and Evaluation of Oculometric Measures in Healthy Participants
Brief Title: A Prospective Study to Evaluate the Correlation Between Oculometric Measurements and Clinical Endpoints in PD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuraLight (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL/PD/2022-1
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Idiopathic Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD patients visiting clinic (Experimental): All patients will undergo a NeuraLight session for oculometric evaluation along with eye-tracking recordings. All assessments will be performed during a clinic visit unless authorized to be conducted remotely.
  Interventions: Other: NeuraLight software-based platform
- Healthy subjects (Experimental): All patients will undergo a NeuraLight session for oculometric evaluation along with eye-tracking recordings. All assessments will be performed during a visit unless authorized to be conducted remotely.
  Interventions: Other: NeuraLight software-based platform

INTERVENTIONS:
Other: NeuraLight software-based platform — NeuraLight is an investigational software-based platform that is used for assessment and evaluation of neurological conditions including PD patients

SUMMARY:
This is a prospective study in a cohort of about 500 patients with Idiopathic Parkinson's disease, examined routinely in the neurological outpatient clinic.

This study aims to evaluate the correlation between oculometric measures and clinical endpoints. Subjects will be evaluated following a physician examination.The evaluations will include MDS-UPDRS examination, as well as an oculometric evaluation for eye movements. In addition, 500 healthy subjects will be evaluated.

DETAILED DESCRIPTION:
This is a prospective study in a cohort of patients with idiopathic PD who are visiting the Parkinson's outpatient clinic. The aim of the study is to evaluate the correlation between oculometric measures and MDS-UPDRS score in subjects who meet the inclusion criteria and who provide a signed Informed Consent.

This study is designed to evaluate the correlation between oculometric measures and the Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS). Subjects will be evaluated at their visit to the clinic. The evaluations will include an MDS-UPDRS examination by a certified neurologist and other tests. In addition, all patients will undergo a NeuraLight session for oculometric evaluation along with eye-tracking recordings. All assessments will be performed during a clinic visit unless authorized to be conducted remotely. In addition, 500 healthy subjects will be evaluated, undergoing a NeuraLight session for oculometric evaluation along with eye-tracking recordings.

ELIGIBILITY:
PD patients:

Inclusion Criteria:

* Men and women with idiopathic PD (Hoehn & Yahr scale 1-5)
* Age between 18 and 85 years old
* Normal or corrected vision
* Ability to follow instructions
* Willing and able to sign an informed consent form

Exclusion Criteria:

* Inability to sit for 20 minutes on a chair in a calm manner
* Personal or 1st degree relative history of epilepsy
* Additional neurological diseases
* Drug or alcohol abuse

Healthy subjects:

Inclusion Criteria:

* Age between 18 and 85 years old
* Normal or corrected vision
* Ability to follow instructions
* Willing and able to sign an informed consent form

Exclusion Criteria

* Inability to sit for 20 minutes on a chair in a calm manner
* Personal or 1st degree relative history of epilepsy
* Neurological diseases
* Drug or alcohol abuse

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Correlation between MDS-UPDRS score and its parts with NeuraLight oculometric measurements | 12 months
  The correlation between MDS-UPDRS score and its parts with NeuraLight oculometric measurements (R-Square>0.5, p<0.05) according to the Movement Disorder Society-Sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) at every visit
Feasibility of using NeuraLight system to capture oculometric measures in a cohort of PD patients and healthy subjects | 12 months
  Capturing >50 different oculometric measures in >95% of a cohort of about 1000 patients
Comparison of NeuraLight extracted oculometric measures with a validated eye-tracking system | 12 months
  Relative root mean square error (RMSE) of NeuraLight's extracted oculometric measures compared with retrieved measurements from a validated eye tracking system <0.1

SECONDARY OUTCOMES:
Using the retrieved data of collected NeuraLight oculometric measures for calibration of prediction models of MDS-UPDRS clinical endpoint | 12 months
  Optimization of a feature selection model (Fisher's Linear Discriminant Analysis (LDA)) on NeuraLight oculometric measures used for a logistic regression model of MDS-UPDRS with a relative root mean square error (RMSE) of <0.1

CONTACTS AND LOCATIONS:
Overall Officials: Johnathan Reiner, MD, Principal Investigator — Sackler Faculty of Medicine, Tel Aviv University
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No
There is not plan to share IPD with other researchers

REFERENCES:
- [Background] Anderson TJ, MacAskill MR. Eye movements in patients with neurodegenerative disorders. Nat Rev Neurol. 2013 Feb;9(2):74-85. doi: 10.1038/nrneurol.2012.273. Epub 2013 Jan 22. PMID 23338283
- [Background] Waldthaler J, Tsitsi P, Svenningsson P. Vertical saccades and antisaccades: complementary markers for motor and cognitive impairment in Parkinson's disease. NPJ Parkinsons Dis. 2019 Jun 24;5:11. doi: 10.1038/s41531-019-0083-7. eCollection 2019. PMID 31263745